CLINICAL TRIAL: NCT04925596
Title: Prescription of Benzodiazepines by General Practitioners: Characteristics of Prescribing Trend and Implementation of an Online Educational Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 47/2016/CEFCM
Record Dates: First submitted 2019-04-10; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Anxiety; Prescription Drug Abuse and Dependency
Keywords: Prescribing Patterns; Benzodiazepines; General Practitioners
MeSH Terms: conditions — Anxiety Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): general practitioners randomized to intervention group will be given access to ePrimaPrescribe online program
  Interventions: Behavioral: ePrimaPrescribe online educational program
- Control (Active Comparator): general practitioners randomized to control group will be given access to an online program concerning doctor-patient communication
  Interventions: Behavioral: ComunicaSaudeMental online educational program

INTERVENTIONS:
Behavioral: ePrimaPrescribe online educational program — online training program aiming to change general practitioners' benzodiazepine prescription
  Arms: Intervention
Behavioral: ComunicaSaudeMental online educational program — online training program aiming to improve general practitioners' communication with mentally ill patients
  Arms: Control

SUMMARY:
Portugal has the highest benzodiazepine utilization compared to other European countries. The high utilization of benzodiazepines has been a concern due to reported side effects of long-term use and dependence. Also, these data demonstrate that doctors are possibly choosing an inadequate treatment to manage anxious and depressive syndromes.

This research aims to develop and implement in primary health care units an online educational program, following a cluster randomized study design; to study the impact of this educational program for changing general practitioner's benzodiazepine prescription pattern; to analyze of barriers and facilitators to the implementation of the e-PrimaPrescribe program.

DETAILED DESCRIPTION:
BZD excessive prescription has long been considered a serious mental health concern in many countries. A large number of interventions using different methodologies have been implemented to change BZD prescription pattern at primary health care settings, with limited positive results.

The investigators propose the implementation of an effectiveness-implementation hybrid type 1 intervention. In the study it was developed an online platform, named ePrimaPrescribe, which was delivered using a Digital Behavior Change Intervention(DBCI).

The investigators included all primary health care units from one region in Portugal which were randomly allocated to receive a Digital Behavior Change Intervention (DBCI) in the format of an online platform to reduce BZD prescription (ePrimaPrescribe) or an online platform concerning communication techniques (control).

The investigators primarily aimed to evaluate the effectiveness of the Digital Behavior Change Intervention (DBCI) using as outcome measure the frequency of BZD prescriptions issued per month. Secondarily the investigators aimed to analyze the effect of ePrimaprescribe on antidepressant prescriptions, to study the effect of ePrimaprescribe on diagnosis definition associated with BZD and antidepressant prescription; to perform a cost analysis considering the monthly National Health Service spending with BZD co-payment. The investigators finally aim to analyze the implementation process using quantitative and qualitative methods.

ELIGIBILITY:
Inclusion Criteria:

* Primary care units using the Portuguese online prescription tool (created by the Portuguese Shared Services of the Ministry of Health and Finance - SPMS)

Exclusion Criteria:

* Primary care units involved in another trial concerning mental health topics directly related with the subject of this thesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2019-04-09 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of BZD prescriptions issued per month | Change from baseline prescription to 6 months after intervention
  Each prescription data was coded using an individual GP and patient numerical identification, in a secured and validated electronic database, directly extracted by the central Shared Services of the Portuguese Ministry of Health.

SECONDARY OUTCOMES:
Change in the frequency of antidepressant prescriptions issued per month | Change from baseline prescription to 6 months after intervention
  Each prescription data was coded using an individual GP and patient numerical identification, in a secured and validated electronic database, directly extracted by the central Shared Services of the Portuguese Ministry of Health.
Change in the diagnosis registration frequency | Change from baseline prescription to 6 months after intervention
  Monthly registration distribution of psychological symptoms, complaints, and diagnoses coded at the same month as BZD and antidepressant prescriptions. The GP's diagnosis registration used the International Classification of Primary Care, second edition (ICPC-2) developed and updated by the World Organization of Family Doctors' (WONCA) International Classification Committee (WICC).
Change in the costs with BZD co-payment | Change from baseline prescription to 6 months after intervention
  Cost analysis considering the monthly National Health Service spending with BZD co-payment. This cost was compared with the amount that would need to be spent to comply with needs and solutions suggested when evaluating GP's perceptions of the feasibility and implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Reis, Md, Principal Investigator — Universidade Nova de Lisboa
Locations (1):
- Faculdade Ciências Médicas Universidade Nova de Lisboa - Nova Medical School, Lisbon, Portugal

REFERENCES:
- [Derived] Reis T, Faria I, Serra H, Xavier M. Barriers and facilitators to implementing a continuing medical education intervention in a primary health care setting. BMC Health Serv Res. 2022 May 13;22(1):638. doi: 10.1186/s12913-022-08019-w. PMID 35562695

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04925596/Prot_SAP_000.pdf